CLINICAL TRIAL: NCT01966133
Title: Randomised Controlled Trial on Adjuvant Transarterial Chemoembolisation After Curative Hepatectomy for Hepatocellular Carcinoma
Brief Title: TACE as an Adjuvant Therapy After Hepatectomy for HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jia Fan (Other)
Responsible Party: Sponsor-Investigator, Jia Fan, President of zhongshan hospital, Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LCI-125-009
Record Dates: First submitted 2013-10-16; First posted 2013-10-21 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Randomised controlled trial; TACE; Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ethiodized Oil; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): no interventions were assigned
- TACE('Ethiodized Oil + Doxorubicin) (Active Comparator): TACE using Ethiodized Oil + Doxorubicin mixture was infused through catheter placed at hepatic artery followed by gelfoam embolisation. This is performed 4-6 weeks after surgery.
  Interventions: Drug: Ethiodized Oil + Doxorubicin

INTERVENTIONS:
Drug: Ethiodized Oil + Doxorubicin — TACE using doxorubicin-lipiodol mixture
  Other Names: doxorubicin-lipiodol mixture
  Arms: TACE('Ethiodized Oil + Doxorubicin)

SUMMARY:
Investigators hypothesise that the use of transarterial chemoembolisation (TACE) after liver resection in patients with hepatocellular carcinoma can eradicate residual cancer cells in the liver and thus improve survival of patients with high risk factors for residual tumor. The aim of this study is to compare the survival of patients with high risk factors for residual tumor undergoing liver resection plus post-operative TACE versus liver resection alone.

DETAILED DESCRIPTION:
Liver resection is the mainstay of curative treatment for hepatocellular carcinoma (HCC). However, recurrence is common after surgery and most occurs in the liver, especially for the patients with high risk factors for residual tumor, such as tumors with a diameter more than 5 cm, multiple nodules, and microvascular invasion. Transarterial chemoembolisation (TACE) is an effective palliative treatment for HCC. It involves the infusion of chemotherapeutic agent admixed with iodised oil followed by embolisation of the hepatic arterial flow using small particles. This procedures allows application of smaller dose of chemotherapy concentrated to the liver and thus is well tolerated with minimal side effects. The main complications of TACE are liver function damage, mild feverish symptoms, vomit , etc. But most of them are reversible.

We conduct a randomised controlled trial evaluating the efficacy of using TACE after hepatectomy in HCC patients with high risk factors for residual tumor (tumors with a diameter more than 5 cm, multiple nodules, or microvascular invasion).

ELIGIBILITY:
Inclusion Criteria:

* HCC patients received curative hepatectomy with negative resection margin
* Tumors with a diameter more than 5 cm, multiple nodules, or microvascular invasion were defined as high risk factors for residual tumor and used for patient stratification.
* Age from 18 to 70
* Child-Pugh class A
* ASA class I to III
* ECOG performance status Grade 0 or 1

Exclusion Criteria:

* Patients receiving concomitant local ablation or previous TACE
* Main portal vein tumour thrombus extraction during hepatectomy
* Tumour arising from caudate lobe
* Presence of extra-hepatic disease
* Impaired liver function with either clinically detected ascites, hepatic encephalopathy, serum albumin < 25g/L or bilirubin > 50micromol/L
* Renal impairment with creatinine > 200micromol/L
* Severe concurrent medical illness persisting > 6 weeks after hepatectomy
* History of other cancer
* Hepatic artery anomaly making TACE not possible
* Allergy to doxorubicin or lipiodol
* Pregnant woman
* Informed consent not available

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-08; Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years after operation

SECONDARY OUTCOMES:
Overall Survival | 3-year after surgery
Complications of transarterial chemoembolisation | 3-month after transarterial chemoembolisation

OTHER OUTCOMES:
Health-related quality of life assessment | 1-year after surgery
  The quality of life assessment was measured by Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire (Chinese version 3)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, Principal Investigator — Liver cancer institute, Fudan university; Jian Zhou, MD, Study Director — Liver Cancer Institute, Zhong Shan Hospital, Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China